CLINICAL TRIAL: NCT01187186
Title: A Phase 1, Open-Label, Single-Dose Study to Assess the Effect of Hepatic Function on the Pharmacokinetics and Safety of ASP1941
Brief Title: A Study to Assess the Effect of Hepatic Function on the Pharmacokinetics and Safety of ASP1941
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sr Manager Clinical Trials Registry, Astellas Pharma Global Development
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 1941-CL-0063
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Liver Disease
Keywords: Liver disease; ASP1941
MeSH Terms: conditions — Liver Diseases | interventions — ipragliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate Hepatic Impairment (Experimental): Subjects with Moderate Hepatic Impairment
  Interventions: Drug: ASP1941
- Normal Hepatic Function (Experimental): Subjects with Normal Hepatic Function
  Interventions: Drug: ASP1941

INTERVENTIONS:
Drug: ASP1941 — oral

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) and safety following oral administration of ASP1941 in subjects with moderate hepatic impairment and in subjects with normal hepatic function based on the Child-Pugh Classification (CPC).

DETAILED DESCRIPTION:
Study drug will be orally administered on Day 1. Subjects will be admitted to the clinic until completion of clinic discharge procedures on Day 7 with an outpatient follow-up visit 6-9 days after clinic discharge.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Moderate Hepatic Impairment

  * Agrees to practice highly effective birth control until 7 days post dose. If female, two years post-menopausal, surgically sterile, and not pregnant or lactating
  * Weights at least 45 kg
  * Body mass index between 18 and 34 kg/m2
  * Meets criteria for moderate hepatic impairment defined by Child-Pugh method
* Subjects with Normal Hepatic Function

  * Agrees to practice highly effective birth control until 7 days post dose. If female, two years post-menopausal, surgically sterile, and not pregnant or lactating
  * Weights at least 45 kg
  * Body mass index between 18 and 34 kg/m2
  * Must have normal hepatic function defined by Child-Pugh method

Exclusion Criteria:

* Subjects with Moderate Hepatic Impairment

  * Has history or presence of biliary obstruction or biliary disease, hepatic encephalopathy, advanced ascites, portal hypertension, esophageal /gastric variceal bleeding, hepatocellular carcinoma, previous liver transplantation.
  * Has severe or moderate renal dysfunction
  * Known to be human immunodeficiency virus (HIV) positive
  * Has clinically significant history or presence of illness, malignancy or immunodeficiency
  * Has had a blood transfusion or donated / lost 450 mL of blood or more within 60 days of study drug administrations or donated plasma within 7 days prior to clinical check-in
  * Has history of alcoholism or drug/chemical/substance abuse within past 2 years
* Subjects with Normal Hepatic Function

  * Has severe or moderate renal dysfunction
  * Known to be human immunodeficiency virus (HIV) positive
  * Has clinically significant history or presence of illness, malignancy or immunodeficiency
  * Has had a blood transfusion or donated / lost 450 mL of blood or more within 60 days of study drug administrations or donated plasma within 7 days prior to clinical check-in
  * Has history of alcoholism or drug/chemical/substance abuse within past 2 years

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables used to assess the effect of hepatic function through analysis of blood samples | 7 days following study drug administration

SECONDARY OUTCOMES:
Pharmacokinetic variables used to assess the effect of hepatic impairment through analysis of blood and urine samples | 7 days following study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (1):
- Miami, Florida, United States